CLINICAL TRIAL: NCT03916484
Title: Piloting a Sequential Multiple-Assignment Randomization Trial to Evaluate AllyQuest: an mHealth Intervention for HIV-positive Young MSM and TWSM to Optimize HIV Medication Adherence and Care Outcomes
Brief Title: AllyQuest Adherence App Intervention for HIV-positive Men Who Have Sex With Men and Transgender Women: Pilot Trial
Acronym: AQ2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Medical University of South Carolina (Other); Wayne State University (Other); Rutgers University (Other); University of Alabama at Birmingham (Other); North Carolina State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-2061; 1R34MH118058-01 (NIH)
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-03

CONDITIONS: Hiv; HIV/AIDS; Medication Adherence; Sexual Behavior; Sexually Transmitted Infections (Not HIV or Hepatitis)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence; Sexual Behavior; Sexually Transmitted Diseases; Hepatitis

STUDY DESIGN:
Intervention Model Description: Sequential multiple assignment randomized trials (SMART) are adaptive interventions. An adaptive intervention is a sequence of decision rules that specify how the intensity or type of treatment should change depending on the patient's needs rather than applying a "one size fits all" approach. The type or dose of the intervention is adjusted based on participant characteristics or response. SMARTs are an efficient and rigorous way to maximize clinical utility and real-world applicability. In this SMART, participants are initially randomized to medication adherence support with one of two intervention approaches (AQ or AQ+NSC). At 3 months, based on protocol defined intervention responsiveness, participants are re-randomized or reassigned to continue their initial intervention approach or to change to the other intervention approach for months 4 - 6 of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AQ HIV Medication Adherence app-delivered intervention (Experimental): AQ: At minimum, intended app usage (dose) is for participant to complete a set of activities (record medication taking, complete a challenge, complete a forum post) one time per day (frequency) for 6 months (duration). The participant may or may not stay solely on AQ throughout the study.
  Interventions: Behavioral: AllyQuest HIV Medication Adherence app-delivered intervention
- AQ HIV Medication Adherence app-delivered intervention + NSC (Experimental): AQ+NSC: At minimum, intended app usage (dose) is for participant to complete a set of activities (record medication taking, complete a challenge, complete a forum post) one time per day (frequency) for 6 months (duration). NSC sessions are scheduled approximately every other week (frequency) and last approximately 30 minutes per session (dose). The participant may or may not stay on AQ+NSC throughout the study.
  Interventions: Behavioral: AllyQuest HIV Medication Adherence app-delivered intervention + NSC
- AQ followed by AQ+NSC (Experimental): At 3 months, those who were initially randomized to AQ who meet protocol defined definition for intervention non-responsiveness, are reassigned to AQ+NSC to complete months 4 - 6 of the trial.
  Interventions: Behavioral: AllyQuest HIV Medication Adherence app-delivered intervention; Behavioral: AllyQuest HIV Medication Adherence app-delivered intervention + NSC
- AQ+NSC followed by AQ (Experimental): At 3 months, those who were initially randomized to AQ+NSC who meet protocol defined definition for intervention responsiveness, may get re-randomized to AQ alone to complete months 4 - 6 of the trial.
  Interventions: Behavioral: AllyQuest HIV Medication Adherence app-delivered intervention; Behavioral: AllyQuest HIV Medication Adherence app-delivered intervention + NSC

INTERVENTIONS:
Behavioral: AllyQuest HIV Medication Adherence app-delivered intervention — AQ provides daily ART reminders and calendar; weekly tailored message; monthly appointment and refill reminders; social support via daily chat wall; daily challenge featuring skills-building and articles; education center; narrative collections; in app "account" rewards daily use by adding or subtracting small financial reward dependent on daily app use; personalized profile and avatar. Participants have 24-hour access to all features of the AQ app.
  Other Names: AQ
  Arms: AQ HIV Medication Adherence app-delivered intervention; AQ followed by AQ+NSC; AQ+NSC followed by AQ
Behavioral: AllyQuest HIV Medication Adherence app-delivered intervention + NSC — In AQ+, participants receive all of AQ and have the added ability to text in the app with an adherence counselor, using Next Step Counseling (NSC). NSC is an interactive, client-centered motivational intervention to improve ART adherence. Key components of NSC include: review experiences with adherence, exploration of adherence facilitators and barriers, identification of adherence needs, identification of strategies to meet needs, and development of an adherence action plan. AQ+ includes unprompted check-in messages from the NSC counselor and scheduled in-app NSC sessions approximately every other week.
  Other Names: AQ+
  Arms: AQ HIV Medication Adherence app-delivered intervention + NSC; AQ followed by AQ+NSC; AQ+NSC followed by AQ

SUMMARY:
AllyQuest (AQ) is a theory-informed smart phone application that supports HIV medication adherence for young men who have sex with men and young transgender women who have sex with men (YMSM/YTW) via behavior change, social support, and game-based mechanics. This study aims to evaluate the feasibility and acceptability of AQ and AQ plus medication adherence counseling in a Sequential Multiple Assignment Randomization Trial.

DETAILED DESCRIPTION:
AllyQuest (AQ) is a theory-informed smart phone application that supports HIV medication adherence for young men who have sex with men and young transgender women who have sex with men (YMSM/YTW) via behavior change, social support, and game-based mechanics. This study aims to evaluate the feasibility and acceptability of AQ and AQ plus medication adherence counseling in a Sequential Multiple Assignment Randomization Trial.

AllyQuest (AQ) is a smart phone application for Android and iOS (Apple) that supports HIV medication adherence. Intervention development was guided by health behavior change theories including Social Cognitive Theory (SCT), narrative communication (e.g. storytelling), and the Fogg Behavioral Model (FBM) of persuasive technology. AQ addresses key principles of SCT including: (1) observational learning by doing daily activities; (2) modeling and vicarious experiences (observing and participating in Daily Discussions, exploration of narrative "choose-your-own-adventure" stories); (3) self-efficacy and verbal persuasion from expert sources (multi-media knowledge center, tailored messages) and (4) reinforcements (virtual rewards, financial incentives, achievements). AQ incorporates principles of the FBM including triggers via app notifications and content, increasing ability via knowledge articles and identifying steps toward behavioral goals, and motivation via social support, rewards, goal setting, and achievement.

This study will test AQ and an enhanced version of AQ (AQ+) that adds two-way text based Next Step Counseling (NSC) for medication adherence. A sequential multiple assignment randomized trial (SMART) is a study design suited to development of adaptive interventions. An adaptive intervention is a sequence of decision rules that specify how the intensity or type of treatment should change depending on the patient's needs rather than applying a "one size fits all" approach. In a SMART, participants are randomized to an initial treatment, and, depending on how they respond, may be assigned or randomized to a new type or intensity of treatment. SMARTs are an efficient and rigorous way to study how the type or dose of treatment should be adjusted based on subject characteristics or response and thus maximize clinical utility and real-world applicability. In this SMART, participants are initially randomized to medication adherence support with one of two intervention approaches (AQ or AQ+NSC). At 3 months, based on protocol defined intervention responsiveness, participants are re-randomized or reassigned to continue their initial intervention approach or to change to the other intervention approach for months 4 - 6 of the trial.

Participants will complete viral load (VL) and web-based computer assisted survey instrument (CASI) assessments at baseline and 3- and 6- months. A sample of 20-25 users will complete a qualitative exit interview to evaluate their experience using AQ and AQ+ and their experience with the escalation/de-escalation intervention strategies.

The study will assess intervention feasibility, acceptability, and preliminary efficacy including: 1) frequency and total time spent on each AQ feature; 2) in-app daily adherence reports; and 3) user-contributed content (adherence counseling chat logs, user-entered daily discussion content and adherence strategies). Analyses will determine which treatment strategies embedded in the SMART (escalation, de-escalation, and maintenance combinations) result in sustained intervention app engagement, self-reported adherence, and viral suppression.

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV
* Assigned male at birth
* currently identify as male or transgender woman
* anal sex with another male or transgender woman(lifetime)
* access to a smart phone with data plan
* English literacy
* prescribed ART
* At least one of the following: Having failed to show up for or missed 1 or more scheduled HIV care appointment in the past 12 months OR Last HIV care visit was more than 6 months ago OR Self-reporting less than 90% ART adherence in the past 4 weeks OR have a detectable viral load measure in the past 12 months OR recently diagnosed with HIV (past 3 months)

Exclusion Criteria:

* younger than 15, or older than 29
* assigned female at birth
* HIV negative or status unknown

Ages: 15 Years to 29 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — The study will enroll self identified men and transgender women.
Enrollment: 71 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Muessig, PhD, Principal Investigator — UNC-Chapel Hill; Lisa Hightow-Weidman, MD, MPH, Principal Investigator — UNC-Chapel Hill
Locations (6):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - Wayne State University, Detroit, Michigan
  - Rutgers University, Newark, New Jersey
  - UNC-Chapel Hill, Chapel Hill, North Carolina
  - RAIN, Charlotte, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 6 clinical recruitment sites in Birmingham, AL; Chapel Hill and Charlotte, NC; Charleston, SC; Detroit, MI and Newark, NJ.
Pre-assignment Details: Enrollment and randomization to stage 1 interventions took place directly following confirmation of eligibility and completion of informed consent. All enrolled participants were randomized and assigned to a stage 1 intervention condition.
Groups:
- AQ HIV Medication Adherence App-delivered Intervention: Participants in this arm received the intervention approach starting with AQ for the first 3 months and remaining with AQ for months 4 - 6.
  AllyQuest HIV Medication Adherence app-delivered intervention: AQ provides daily ART reminders and calendar; weekly tailored message; monthly appointment and refill reminders; social support via daily chat wall; daily challenge featuring skills-building and articles; education center; narrative collections; in app "account" rewards daily use by adding or subtracting small financial reward dependent on daily app use; personalized profile and avatar. Participants have 24-hour access to all features of the AQ app.
- AQ HIV Medication Adherence App-delivered Intervention + NSC: Participants in this arm received the intervention approach starting with AQ+NSC for the first 3 months and remaining with AQ+NSC for months 4 - 6.
  AllyQuest HIV Medication Adherence app-delivered intervention + NSC: In AQ+, participants receive all of AQ and have the added ability to text in the app with an adherence counselor, using Next Step Counseling (NSC). NSC is an interactive, client-centered motivational intervention to improve ART adherence. Key components of NSC include: review experiences with adherence, exploration of adherence facilitators and barriers, identification of adherence needs, identification of strategies to meet needs, and development of an adherence action plan. AQ+ includes unprompted check-in messages from the NSC counselor and scheduled in-app NSC sessions approximately every other week.
- AQ Followed by AQ+NSC: Participants in this arm received the intervention approach starting with AQ for the first 3 months and escalated to AQ+NSC for months 4 - 6, having met the protocol definition for intervention non-responsiveness.
  AllyQuest HIV Medication Adherence app-delivered intervention: AQ provides daily ART reminders and calendar; weekly tailored message; monthly appointment and refill reminders; social support via daily chat wall; daily challenge featuring skills-building and articles; education center; narrative collections; in app "account" rewards daily use by adding or subtracting small financial reward dependent on daily app use; personalized profile and avatar. Participants have 24-hour access to all features of the AQ app.
  AllyQuest HIV Medication Adherence app-delivered intervention + NSC: In AQ+, participants receive all of AQ and have the added ability to text in the app with an adherence counselor, using Next Step Counseling (NSC). NSC is an interactive, client-centered motivational intervention to improve ART adherence. Key components of NSC include: review experiences with adherence, exploration of adherence facilitators and barriers, identification of adherence needs, identification of strategies to meet needs, and development of an adherence action plan. AQ+ includes unprompted check-in messages from the NSC counselor and scheduled in-app NSC sessions approximately every other week.
- AQ+NSC Followed by AQ: Participants in this arm received the intervention approach starting with AQ+NSC for the first 3 months and de-escalated to AQ for months 4 - 6, having met the protocol definition for intervention responsiveness.
  AllyQuest HIV Medication Adherence app-delivered intervention: AQ provides daily ART reminders and calendar; weekly tailored message; monthly appointment and refill reminders; social support via daily chat wall; daily challenge featuring skills-building and articles; education center; narrative collections; in app "account" rewards daily use by adding or subtracting small financial reward dependent on daily app use; personalized profile and avatar. Participants have 24-hour access to all features of the AQ app.
  AllyQuest HIV Medication Adherence app-delivered intervention + NSC: In AQ+, participants receive all of AQ and have the added ability to text in the app with an adherence counselor, using Next Step Counseling (NSC). NSC is an interactive, client-centered motivational intervention to improve ART adherence. Key components of NSC include: review experiences with adherence, exploration of adherence facilitators and barriers, identification of adherence needs, identification of strategies to meet needs, and development of an adherence action plan. AQ+ includes unprompted check-in messages from the NSC counselor and scheduled in-app NSC sessions approximately every other week.
Period: Stage 1 Intervention (Months 1-3)
Arm/Group | AQ HIV Medication Adherence App-delivered Intervention | AQ HIV Medication Adherence App-delivered Intervention + NSC | AQ Followed by AQ+NSC | AQ+NSC Followed by AQ
Started | 7 | 41 | 15 | 8
Completed | 7 | 40 | 15 | 8
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: Stage 2 Intervention (Months 4-6)
Arm/Group | AQ HIV Medication Adherence App-delivered Intervention | AQ HIV Medication Adherence App-delivered Intervention + NSC | AQ Followed by AQ+NSC | AQ+NSC Followed by AQ
Started | 7 | 40 | 15 | 8
Completed | 5 | 29 | 11 | 7
Not Completed | 2 | 11 | 4 | 1
Not completed — Lost to Follow-up | 2 | 11 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- AQ HIV Medication Adherence App-delivered Intervention: Participants in this arm received the intervention approach starting with AQ for the first 3 months and remaining with AQ for months 4 - 6.
- AQ HIV Medication Adherence App-delivered Intervention + NSC: Participants in this arm received the intervention approach starting with AQ+NSC for the first 3 months and remaining with AQ+NSC for months 4 - 6.
- AQ Followed by AQ+NSC: Participants in this arm received the intervention approach starting with AQ for the first 3 months and escalated to AQ+NSC for months 4 - 6, having met the protocol definition for intervention non-responsiveness.
- AQ+NSC Followed by AQ: Participants in this arm received the intervention approach starting with AQ+NSC for the first 3 months and de-escalated to AQ for months 4 - 6, having met the protocol definition for intervention responsiveness.
- Total: Total of all reporting groups
Arm/Group | AQ HIV Medication Adherence App-delivered Intervention | AQ HIV Medication Adherence App-delivered Intervention + NSC | AQ Followed by AQ+NSC | AQ+NSC Followed by AQ | Total
Number analyzed (Participants) | 7 | 41 | 15 | 8 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 1 | 0 | 4
  Between 18 and 65 years | 6 | 39 | 14 | 8 | 67
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 24.28 [16 to 29] | 22.43 [18 to 28] | 22.13 [18 to 28] | 22.37 [19 to 27] | 22.54 [16 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 7 | 41 | 15 | 8 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 2 | 0 | 8
  Not Hispanic or Latino | 6 | 35 | 13 | 8 | 62
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 2
  Black or African American | 6 | 27 | 8 | 8 | 49
  White | 1 | 3 | 2 | 0 | 6
  More than one race | 0 | 8 | 5 | 0 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 41 | 15 | 8 | 71
Mean Percent of Past 30-Day ART medication adherence [Mean (Standard Deviation); unit: percentage of doses taken] — HIV Antiretroviral (ART) Medication Adherence is measured by computer-assisted self interview (CASI) as percent of prescribed ART doses taken in the past 30 days. Population: This survey question was optional for participants. The number analyzed includes all participants who answered this question.
  percentage of doses taken
    number analyzed (Participants) | 5 | 35 | 11 | 8 | 59
    (all) | 98.00 (2.73) | 81.05 (28.37) | 78.09 (28.59) | 94.00 (12.67) | 83.69 (25.98)
Participants with viral suppression [Count of Participants; unit: Participants] — Viral suppression is defined as having an HIV viral load below the lower limit of detection per assay used.
  Participants | 2 | 14 | 8 | 5 | 29

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility: Average Proportion of Days of Any App Use
Description: The average proportion of days of any app use during the trial across all participants as recorded by the app backend para data. Total possible range: 0 - 1. Higher proportion indicates higher intervention feasibility.
Time Frame: 180 days
Population: Per the pre-specified analysis plan, this outcome compares how effective each intervention sequence performed as measured by participants' daily use of the intervention app with the 4 sequences offering different intervention intensity variations.
Measure: Mean (Standard Deviation); unit: proportion of days
Groups:
- Total Sample: All enrolled participants
Arm/Group | AQ HIV Medication Adherence App-delivered Intervention | AQ HIV Medication Adherence App-delivered Intervention + NSC | AQ Followed by AQ+NSC | AQ+NSC Followed by AQ | Total Sample
Number analyzed (Participants) | 7 | 41 | 15 | 8 | 71
proportion of days | 0.64 (0.17) | 0.40 (0.33) | 0.27 (0.14) | 0.64 (0.16) | 0.42 (0.29)

2. Primary Outcome: Intervention Feasibility: Average Proportion of Days of HIV Medication Tracked
Description: The average proportion of days participants used the app to track their HIV medication taking. Total possible range: 0 - 1. Higher proportion indicates higher intervention feasibility.
Time Frame: 180 Days
Population: Per the pre-specified analysis plan, this outcome compares how effective each intervention sequence performed as measured by participants' daily use of the intervention app to track daily medication with the 4 sequences offering different intervention intensity variations.
Measure: Mean (Standard Deviation); unit: proportion of days
Groups:
- Total Sample: This group includes all enrolled participants
Arm/Group | AQ HIV Medication Adherence App-delivered Intervention | AQ HIV Medication Adherence App-delivered Intervention + NSC | AQ Followed by AQ+NSC | AQ+NSC Followed by AQ | Total Sample
Number analyzed (Participants) | 7 | 41 | 15 | 8 | 71
proportion of days | 0.80 (0.15) | 0.50 (0.33) | 0.38 (0.20) | 0.81 (0.13) | 0.54 (0.31)

3. Primary Outcome: Intervention Acceptability: Mean Intervention Acceptability CSQ-8 Score
Description: The mean composite score calculated from the Client Satisfaction Questionnaire (CSQ-8), an 8-item validated scale measuring the construct of global intervention satisfaction. Total possible composite score range: 8 (lowest acceptability, worst outcome) to 32 (highest acceptable, best outcome).
Time Frame: 6 Months
Population: The protocol was amended to utilize a more precise scale for this measure (see outcome #4). The CSQ-8® was not administered and no data were collected using this tool.
Arm/Group | AQ HIV Medication Adherence App-delivered Intervention | AQ HIV Medication Adherence App-delivered Intervention + NSC | AQ Followed by AQ+NSC | AQ+NSC Followed by AQ
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Primary Outcome: Intervention Acceptability: Mean Intervention Acceptability Score
Description: The mean composite score is calculated from the Acceptability of Health Apps among Adolescents (AHAA) scale, a 22-item validated scale measuring the construct of global intervention acceptability. Item response options include: Strongly Disagree, Disagree, Agree, Strongly Agree. Scale items are grouped into 6 sub-scales. Responses to the items in each sub-scale are averaged and the sub-scale averages are added to obtain a total possible composite score ranging from 6 (lowest acceptability, worst outcome) to 24 (highest acceptable, best outcome). A score of 18 or higher is consistent with overall high acceptability.
Time Frame: 6 Months
Population: Participants could choose to decline to answer some or all of the self-reported CASI responses to intervention acceptability measures. This analysis includes all participants who answered half or more (>=11) of the 22 items on the AHAA scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AQ HIV Medication Adherence App-delivered Intervention | AQ HIV Medication Adherence App-delivered Intervention + NSC | AQ Followed by AQ+NSC | AQ+NSC Followed by AQ | Total Sample
Number analyzed (Participants) | 6 | 28 | 7 | 6 | 47
score on a scale | 20.95 (1.37) | 19.97 (2.32) | 18.36 (0.61) | 17.06 (4.23) | 19.48 (2.60)

5. Secondary Outcome: Mean Percent of Past 30-Day ART Medication Adherence
Description: HIV Antiretroviral (ART) Medication Adherence is measured by CASI as percent of ART doses taken in the past 30 days.
Time Frame: Month 6 follow-up time point
Population: Data are reported for all participants who completed this question on the 6-month follow-up survey
Measure: Mean (Standard Deviation); unit: percentage of doses taken
Arm/Group | AQ HIV Medication Adherence App-delivered Intervention | AQ HIV Medication Adherence App-delivered Intervention + NSC | AQ Followed by AQ+NSC | AQ+NSC Followed by AQ | Total Sample
Number analyzed (Participants) | 5 | 20 | 11 | 7 | 43
percentage of doses taken | 99.00 (1.73) | 88.15 (22.47) | 97.09 (4.32) | 84.42 (25.35) | 91.09 (18.80)
Statistical Analysis 1: Comparison: AQ HIV Medication Adherence App-delivered Intervention vs AQ HIV Medication Adherence App-delivered Intervention + NSC vs AQ Followed by AQ+NSC vs AQ+NSC Followed by AQ; Test type: Other; p = 0.33, Kruskal-Wallis — No a priori threshold for statistical significance was specified

6. Secondary Outcome: Mean Percent ART Medication Adherence Over Time
Description: HIV Antiretroviral (ART) Medication Adherence is measured by CASI as percent of prescribed ART doses taken in the past 30 days. Assessed at Baseline and Month 6 follow-up time point.
Time Frame: up to 6 months
Population: Analysis population includes all those who answered this question on both the Baseline and the Month 6 follow-up surveys.
Measure: Mean (Standard Deviation); unit: percentage of medication taken
Arm/Group | AQ HIV Medication Adherence App-delivered Intervention | AQ HIV Medication Adherence App-delivered Intervention + NSC | AQ Followed by AQ+NSC | AQ+NSC Followed by AQ | Total Sample
Number analyzed (Participants) | 4 | 18 | 7 | 7 | 36
percentage of medication taken
  Baseline | 98.75 (2.50) | 80.77 (31.10) | 73.00 (32.34) | 98.42 (2.07) | 84.69 (27.31)
  Month 6 Follow-up | 98.75 (1.89) | 87.16 (23.53) | 96.85 (5.17) | 84.42 (25.35) | 89.80 (20.31)
Statistical Analysis 1: Comparison: AQ HIV Medication Adherence App-delivered Intervention; Test type: Other; p = 1.00, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: AQ HIV Medication Adherence App-delivered Intervention + NSC; Test type: Other; p = 0.43, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: AQ Followed by AQ+NSC; Test type: Other; p = 0.06, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: AQ+NSC Followed by AQ; Test type: Other; p = 0.06, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Total Sample; Test type: Other; p = 0.48, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Number of Participants With Viral Suppression
Description: Viral suppression is defined as having an HIV viral load below the lower limit of detection per assay used. The study will report the number of participants who are virally suppressed at 6 month follow-up.
Time Frame: Month 6 follow-up time point
Population: All participants with an available viral load lab measure for the 6-month follow-up time point.
Measure: Count of Participants; unit: Participants
Arm/Group | AQ HIV Medication Adherence App-delivered Intervention | AQ HIV Medication Adherence App-delivered Intervention + NSC | AQ Followed by AQ+NSC | AQ+NSC Followed by AQ | Total Sample
Number analyzed (Participants) | 5 | 25 | 11 | 7 | 48
Participants | 3 | 19 | 8 | 3 | 33
Statistical Analysis 1: Comparison: AQ HIV Medication Adherence App-delivered Intervention vs AQ HIV Medication Adherence App-delivered Intervention + NSC vs AQ Followed by AQ+NSC vs AQ+NSC Followed by AQ; Test type: Other; p = 0.45, Fisher Exact — No a priori threshold for statistical significance was specified

8. Secondary Outcome: Percent of Participants With Viral Suppression Over Time
Description: Viral suppression is defined as having an HIV viral load below the lower limit of detection per assay used. Assessed at Baseline and Month 3 follow-up time point.
Time Frame: up to 3 months
Population: Includes all participants who had available clinical viral load measures at both baseline and month 3 follow-up. This outcome reports on viral suppression at the end of Stage 1 of the intervention (Month 3 follow-up visit).
Measure: Number; unit: percent of participants
Groups:
- Stage 1: AQ HIV Medication Adherence App-delivered Intervention: Group includes those initially randomized to AQ alone for Months 1 to 3.
- Stage 1: AQ HIV Medication Adherence App-delivered Intervention + NSC: Group includes those initially randomized to AQ+NSC for Months 1 to 3.
Arm/Group | Stage 1: AQ HIV Medication Adherence App-delivered Intervention | Stage 1: AQ HIV Medication Adherence App-delivered Intervention + NSC | Total Sample
Number analyzed (Participants) | 15 | 33 | 48
percent of participants
  Baseline | 40.00 | 33.33 | 35.42
  Month 3 follow-up | 80.00 | 75.76 | 77.08
Statistical Analysis 1: Comparison: Total Sample; Test type: Other; p < 0.001, McNemar
Statistical Analysis 2: Comparison: Stage 1: AQ HIV Medication Adherence App-delivered Intervention; Test type: Other; p = 0.07, McNemar
Statistical Analysis 3: Comparison: Stage 1: AQ HIV Medication Adherence App-delivered Intervention + NSC; Test type: Other; p = 0.003, McNemar

9. Secondary Outcome: Percent of Participants With Viral Suppression Over Time
Description: Viral suppression is defined as having an HIV viral load below the lower limit of detection per assay used. Assessed at Baseline and Month 6 follow-up.
Time Frame: up to 6 months
Population: Population includes all participants with an available clinical viral load measure at both the baseline and month 6 follow-up.
Measure: Number; unit: percent of participants
Arm/Group | AQ HIV Medication Adherence App-delivered Intervention | AQ HIV Medication Adherence App-delivered Intervention + NSC | AQ Followed by AQ+NSC | AQ+NSC Followed by AQ | Total Sample
Number analyzed (Participants) | 5 | 25 | 11 | 7 | 48
percent of participants
  Baseline | 0.00 | 28.00 | 45.45 | 71.43 | 35.42
  Month 6 follow-up | 60.00 | 76.00 | 72.73 | 42.86 | 68.75
Statistical Analysis 1: Comparison: AQ HIV Medication Adherence App-delivered Intervention; Test type: Other; p = 0.25, McNemar
Statistical Analysis 2: Comparison: AQ HIV Medication Adherence App-delivered Intervention + NSC; Test type: Other; p = 0.002, McNemar
Statistical Analysis 3: Comparison: AQ Followed by AQ+NSC; Test type: Other; p = 0.453, McNemar
Statistical Analysis 4: Comparison: AQ+NSC Followed by AQ; Test type: Other; p = 0.500, McNemar
Statistical Analysis 5: Comparison: Total Sample; Test type: Other; p = 0.003, McNemar

ADVERSE EVENTS:
Time Frame: From time of initial consent through 6-month Follow-Up, a total of approximately 6 months.
Groups:
- Stage 1: (Months 1-3) AQ HIV Medication Adherence App-delivered Intervention: Participants in this arm received the intervention approach starting with AQ for the first 3 months.
- Stage 1: (Months 1-3) AQ+NSC HIV Medication Adherence App-delivered Intervention + NSC: Participants in this arm received the intervention approach starting with AQ+NSC for the first 3 months.
- Stage 2: (Months 4-6) AQ HIV Medication Adherence App-delivered Intervention: Participants in this arm received the intervention approach of AQ for months 4 - 6.
- Stage 2: (Months 4-6) AQ HIV Medication Adherence App-delivered Intervention + NSC: Participants in this arm received the intervention approach of AQ+NSC for months 4 - 6.
Arm/Group | Stage 1: (Months 1-3) AQ HIV Medication Adherence App-delivered Intervention | Stage 1: (Months 1-3) AQ+NSC HIV Medication Adherence App-delivered Intervention + NSC | Stage 2: (Months 4-6) AQ HIV Medication Adherence App-delivered Intervention | Stage 2: (Months 4-6) AQ HIV Medication Adherence App-delivered Intervention + NSC
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/49 | 0/15 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/49 | 0/15 | 0/55
Other Adverse Events (participants affected / at risk) | 0/22 | 0/49 | 0/15 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT03916484/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT03916484/ICF_002.pdf